CLINICAL TRIAL: NCT05306873
Title: A Phase 2, Double-Blind, Placebo-Controlled Trial of Mycophenolate Mofetil Alone or With Voclosporin for Systemic Lupus: Examining Distinct Immunophenotypes to Validate and Enhance Rational Treatment (DIVERT) (ALE10)
Brief Title: Examining Distinct Immunophenotypes to Validate and Enhance Rational Treatment in Systemic Lupus
Acronym: DIVERT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed due to slow enrollment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ALE10
Record Dates: First submitted 2022-03-11; First posted 2022-04-01 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus; Mycophenolate Mofetil; Voclosporin
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Mycophenolic Acid; voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MMF (Experimental): Participants will receive 500 mg mycophenolate mofetil (MMF) bid for 7 days, followed by 500mg and 1,000mg MMF in divided doses for 7 days. They will then continue at a stable dose of 1,000mg MMF bid. Visits to evaluate AEs, vital signs, hematology and chemistry, study medication compliance, medication use, disease status, participant reported outcomes, and to obtain biomarker samples will occur every 4 weeks after randomization
  Interventions: Drug: Mycophenolate Mofetil
- Placebo for MMF (Placebo Comparator): Participants will receive 500 mg corresponding mycophenolate mofetil (MMF) placebo bid for 7 days, followed by 500mg and 1,000mg corresponding MMF placebo in divided doses for 7 days. They will then continue at a stable dose of 1,000mg corresponding MMF placebo bid. Visits to evaluate AEs, vital signs, hematology and chemistry, study medication compliance, medication use, disease status, participant reported outcomes, and to obtain biomarker samples will occur every 4 weeks after randomization
  Interventions: Drug: Placebo for Mycophenolate Mofetil
- MMF+ Placebo for Voclosporin (Experimental): Participants randomized in this arm will receive up to 24 weeks of mycophenolate mofetil (MMF) plus placebo for voclosporin, also during the first 2 weeks of treatment, a single intramuscular injection of a long-acting corticosteroid may be administered if needed to achieve amelioration of symptoms without meeting the definition of treatment failure in Stage 3 and without a requirement to stop Stage 3 study-provided medication
  Interventions: Drug: Placebo for Voclosporin; Drug: Mycophenolate Mofetil
- MMF+ Voclosporin (Experimental): Participants randomized in this arm will receive up to 24 weeks of mycophenolate mofetil (MMF) plus voclosporin, also during the first 2 weeks of treatment, a single intramuscular injection of a long-acting corticosteroid may be administered if needed to achieve amelioration of symptoms without meeting the definition of treatment failure in Stage 3 and without a requirement to stop Stage 3 study-provided medication
  Interventions: Drug: Voclosporin; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Stage 2 Dosing:
  Week 1: Participants will receive 500mg MMF/Placebo twice daily
  Week 2: Participants will receive 500mg/Placebo in the morning and 1,000mg MMF/Placebo in the evening
  Weeks 3-48: Participants will receive 1000mg MMF/Placebo twice daily
  Other Names: CellCept; MMF
  Arms: MMF
Drug: Placebo for Mycophenolate Mofetil — Stage 2 Dosing:
  Week 1: Participants will receive 500mg MMF/Placebo twice daily Week 2: Participants will receive 500mg/Placebo in the morning and 1,000mg MMF/Placebo in the evening Weeks 3-48: Participants will receive 1000mg MMF/Placebo twice daily
  Other Names: CellCept; MMF
  Arms: Placebo for MMF
Drug: Voclosporin — Weeks 1-24: 23.7 mg Voclosporin (3 x 7.9 capsules) twice daily
  Other Names: Lupkynis; Lupkynis(TM)
  Arms: MMF+ Voclosporin
Drug: Placebo for Voclosporin — Weeks 1-24: 23.7 mg Placebo for Voclosporin (3 x 7.9 capsules) twice daily
  Arms: MMF+ Placebo for Voclosporin
Drug: Mycophenolate Mofetil — Stage 3 Dosing:
  Participants who received placebo MMF in Stage 2:
  * Week 1: Participants will receive 500mg MMF plus matching placebo for MMF (to appear like a 1000mg dose) twice daily
  * Week 2: Participants will receive 500mg plus matching placebo for MMF (to appear like a 1000mg dose) and 1000mg in divided doses
  * Weeks 3-24: 1000mg MMF twice daily
  Participants who received MMF in Stage 2
  • Week 1-24: 1000mg MMF twice daily
  Other Names: CellCept; MMF
  Arms: MMF+ Placebo for Voclosporin; MMF+ Voclosporin

SUMMARY:
The primary purpose of this study is to evaluate the potential effectiveness of 24 weeks of MMF within previously discovered immunologically defined subsets of SLE patients. Treatment effects will be evaluated within the individual immunologically-homogenous subsets defined at screening. This study will also explore and compare pre-randomization gene expression patterns among responders and non-responders to MMF and MMF plus voclosporin, use comprehensive immunophenotyping to study the immunologic changes that accompany treatment- induced disease improvement and to better understand immunologic changes associated with the loss of clinical response.

DETAILED DESCRIPTION:
The study was conducted in 3 stages with a maximum participant follow-up time of 56 weeks. Stage 1 was a treatment withdrawal period lasting up to 4 weeks where consenting participants receive up to 3 intramuscular injections of a long-acting corticosteroid to achieve amelioration of symptoms. In addition, participants withdraw from all other treatments for lupus with the following exceptions:

(i) as needed (PRN) nonsteroidal anti-inflammatory treatments may be started or continued, (ii) PRN topicals may be continued, (iii) hydroxychloroquine, chloroquine, or quinacrine may be continued at any stable dose, and (iv) prednisone, if<= 10 mg/day, may be continued at stable doses but not started.

Qualifying participants from Stage 1 were randomized (1:1) into Stage 2 to receive either MMF or placebo for MMF for up to 48 weeks. Participants who experienced a Stage 2 treatment failure at or before the Week 24 visit and a corticosteroid injection was deemed sufficient for treatment without new or increased lupus medication were eligible to re-randomize (1:1) into Stage 3 to receive either MMF + Voclosporin or MMF + Placebo for Voclosporin for up to 24 Weeks.

Participants who did not experience a Stage 2 treatment failure at or before the Stage 2 Week 48 visit were to return for an End of Study/Safety Follow-up visit 4 weeks after the final dose of study-provided medication. Similarly, participants who did not experience a Stage 3 treatment failure at or before the Stage 3 Week 24 visits were asked to return for an End of Study/Safety Follow-up visit 4 weeks after the final dose of study provided medication.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be eligible for randomization as study participants.

1. Aged ≥ 18 and ≤ 60 years at the time of informed consent.
2. Meets EULAR/ACR 2019 criteria for SLE.
3. Moderately severe, active, but non-organ threatening disease. Specifically, signs or symptoms meeting criteria for a minimum of:

   1. 1 BILAG A (severe) score in the constitutional, musculoskeletal or mucocutaneous system at the time of screening. See Exclusion Criteria number 2 for additional detail.
   2. 2 BILAG B (moderate) activity scores in any organ systems; or
   3. 1 BILAG B (moderate) activity score in any organ systems and a SELENA-SLEDAI score of ≥ 6.

      * If there is only 1 BILAG B score:

        * If a musculoskeletal BILAG B is scored due to moderate arthritis, where some loss off functional range of movements was present on several days over the last 4 weeks, there must also be a minimum of at least 3 joints that are both tender and swollen due to lupus disease activity in wrists, MCPs or PIPs for the participant to qualify.
        * If a mucocutaneous BILAG B is scored due to acute or subacute cutaneous skin eruption, the rash must cover at least 4% of the body surface area for the participant to qualify. Any active discoid lesion or other form of chronic cutaneous lupus would be qualifying.
4. Approval, by an adjudication committee of a brief entry packet describing the type, severity and duration of symptoms meeting the minimal criteria for entry. The participant will meet this criterion if the committee is confident of all of the following:

   1. Convincing diagnosis of SLE,
   2. Active disease, due to SLE, warranting the potential of dual therapy with potent immune modulators,
   3. No medical or other condition to contraindicate participation in a placebo-controlled, outpatient study of this design.
5. Women of childbearing potential must have a negative serum pregnancy test at screening.
6. Able or willing to use reliable methods of contraception, as outlined in the Mycophenolate REMS brochure for health care providers, from 4 weeks prior to first randomization to 6 weeks after completion of the study. This criterion applies to females of reproductive potential.

   Inclusion Criteria Required Prior to Randomization

   Participants who meet the following criterion at the Stage 2 Randomization Visit may proceed to randomization in Stage 2:
7. After completion of corticosteroid injection(s) and prior to randomization in Stage 2, the participant and his/her physician must agree that disease activity has improved sufficiently from screening such that randomization is acceptable.

   1. The physician must score the CGI-C as "moderately better" or "much better" prior to randomization.

      • The reference value for the CGI-C should be the investigator's determination of the participant's condition at the Screening Visit.
   2. The participant must agree that his/her symptoms have improved (yes/no).

Exclusion Criteria

Participants who meet any of the following criteria are not eligible for randomization as study participants:

1. Inability or unwillingness of a participant to understand and provide written informed consent or comply with the study protocol.
2. BILAG A (severe) disease in the Cardiorespiratory, Neuropsychiatric, Gastrointestinal, Ophthalmic, Renal, or Hematological Systems.
3. Severe or unstable nephritis defined as any of the following:

   1. History of confirmed Class 3-5 nephritis within the last 2 years,
   2. History of confirmed Class 3-5 nephritis > 2 years ago in the absence of documented treatment including both induction and maintenance therapy,
   3. UPCR > 1 g/g at screening, • If UPCR is > 0.5 g/g and ≤ 1 g/g at screening, then a second assessment must be completed with at least 1 week between assessments. If the second assessment is > 1 g/g or has increased by ≥ 0.3 g/g, then the participant is excluded.
4. Evidence of chronic kidney disease defined as eGFR < 45 mL/min per 1.73 m2 at screening, where 175 x (Creatinine/88.4)-1.154 x (Age)-0.203 x (0.742 if female) x (1.212 if of African descent).
5. History of cirrhosis or chronic liver disease unrelated to SLE other than fatty liver disease.
6. History, within 1 year of the Screening Visit, of uncontrolled SLE that would have warranted a BILAG A (except mucocutaneous, constitutional, musculoskeletal) including, but not limited to, hemolytic anemia, neuropsychiatric lupus, or interstitial lung disease.
7. Uncontrolled HTN at the Screening or Randomization Visits defined as a blood pressure > 150/100 with or without treatment, not to exceed 3 complementary antihypertensive treatments.
8. Any of the following laboratory values during screening:

   1. Hemoglobin (Hg) < 8.0 g/dL,
   2. WBC < 2.0 x 10^9 cells/L,
   3. ANC < 1.0 x 10^9 cells/L,
   4. Platelets < 60 x 10^9 cells/L at screening,

      • If platelets < 70 x 10^9 cells/L at screening, platelet count should be retested 2 weeks later. If platelets are < 60 x 10^9 cells/L at retest, participant will be excluded
   5. AST or ALT > 2.5 times the ULN,
   6. Serum IgG levels < 5 g/L
9. Use of ≥ 40 mg/day of prednisone within 4 weeks prior to the Screening Visit or use of > 20 mg/day of prednisone at screening.
10. Unwilling or unable to taper to ≤ 10 mg/day of prednisone or equivalent by the day of randomization.
11. Use of hydroxychloroquine, chloroquine, or quinacrine, if taking, at a prescribed dose that has not been stable for at least 2 months prior to randomization.
12. Use of MMF within 1 year of randomization.
13. Use of CNIs within 3 months of randomization. Topical formulations applied stably for at least one month are allowed.
14. Use of rituximab, obinutuzumab, ocrelizumab, or long-acting B cell depletion agents within 1 year of randomization. Use of agents ≥ 6 months and within 1 year of randomization is permitted if there is evidence of B cell reconstitution as defined as CD19+ counts of ≥ 50 cells/µL.
15. History of intolerance or allergy to MMF, voclosporin, or long-acting corticosteroid preparations.
16. Individuals with known hypersensitivity to Polysorbate 80 (Tween).
17. A woman who is pregnant, breastfeeding, or planning pregnancy from the time of consent until 6 weeks after completion of the study.
18. Any participant with plans for major surgery during the time of the trial.
19. Active infections requiring hospitalization or intravenous antibiotics within 1 month prior to the Screening Visit.
20. Any grade 2 infection or higher from 14 days prior to the Screening Visit and through the screening period that has not resolved by randomization.
21. Acute herpes zoster within 4 months of the Screening Visit.
22. Positive results from a SARS-CoV-2 antigen test administered 2 days prior to and on the day of first randomization.
23. Positive Quantiferon Gold (or equivalent) assay. Indeterminate Quantiferon Gold (or equivalent) assays must be repeated (with same or other interferon gamma release assay per local policy) and shown to be negative. Alternatively, if the Quantiferon Gold (or equivalent) assay remains indeterminate, a participant must have a negative PPD. Finally, if the participant has had the BCG vaccine or has some other condition complicating the interpretation of TB testing, consultation with infection disease specialist must be obtained.

    • Participants diagnosed with latent TB are eligible but must have received appropriate prophylaxis for 30 days prior to initiation of Stage 2 treatment.
24. Serologic evidence at screening of chronic infections including:

    1. HIV infection.
    2. Hepatitis B as indicated by surface antigen or hepatitis B core antibody positivity; if a participant has an isolated positive hepatitis B core antibody, they will be eligible to participate in the study if they are negative for reflex viral load at Screening.
    3. Hepatitis C as indicated by anti-hepatitis C antibody positivity; if a participant is Hepatitis C antibody positive, they will be eligible to participate in the study if they are negative for viral load at Screening.
25. Current, diagnosed, or self-reported drug or alcohol abuse within the last 6 months that, in the opinion of the investigator, would interfere with the ability to comply with study protocol.
26. Recipient of live attenuated vaccine(s) within 8 weeks of the Screening Visit.
27. Use of investigational drugs (excluding SARS-CoV-2 vaccinations or SARS-CoV2 therapeutics) within 8 weeks of the Screening Visit or 5 half-lives, whichever is longer.
28. Past or current mental or physical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Merrill, M.D., Study Chair — Oklahoma Medical Research Foundation: Arthritis and Clinical Immunology Research Program
Locations (10):
- United States (10):
  - UCLA Medical Center: Division of Rheumatology, Los Angeles, California
  - Yale University School of Medicine: Rheumatology, Allergy & Immunology, New Haven, Connecticut
  - Emory University School of Medicine: Division of Rheumatology, Atlanta, Georgia
  - Piedmont Healthcare: Rheumatology Atlanta, Atlanta, Georgia
  - Massachusetts General Hospital: Rheumatology, Allergy and Immunology, Center for Immunology and Inflammatory Diseases, Boston, Massachusetts
  - Feinstein Institute for Medical Research: Center for Autoimmune and Musculoskeletal Diseases, Manhasset, New York
  - Columbia University Medical Center: Department of Medicine, Division of Rheumatology, New York, New York
  - University of North Carolina at Chapel Hill; Thurston Arthritis Research Center: Division of Rheumatology, Allergy, and Immunology, Chapel Hill, North Carolina
  - Oklahoma Medical Research Foundation: Arthritis and Clinical Immunology Research Program, Oklahoma City, Oklahoma
  - PennState Health Milton S. Hershey Medical Center: Division of Rheumatology, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: Autoimmunity Centers of Excellence — https://www.autoimmunitycenters.org/
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 sites were activated in the United States, beginning in October 2022. In Stage 1, 12 consenting participants received an intramuscular injection of a long-acting corticosteroid injection and withdrew from all other treatments for lupus. In Stage 2, 8 eligible participants were randomized to receive either MMF or placebo. In Stage 3, 3 eligible participants from Stage 2 were re-randomized to receive either MMF + Voclosporin or MMF + Placebo.
Pre-assignment Details: A total of 12 participants consented from November 2022 to April 2024 at 7 sites.
Groups:
- Stage 2 MMF: Participants receive up to 48 weeks of MMF. A scheduled ramp-up takes place for the first two weeks. Participants receive 500 mg of MMF twice a day for 7 days, followed by 500 mg and 1000 mg of MMF in divided doses for 7 days, followed by a continued stable dose of 1000 mg of MMF twice a day.
- Stage 2 Placebo for MMF: Participants receive up to 48 weeks of placebo for MMF. A scheduled ramp-up takes place for the first two weeks. Participants receive 500 mg of placebo twice a day for 7 days, followed by 500 mg and 1000 mg of placebo in divided doses for 7 days, followed by a continued stable dose of 1000 mg of placebo twice a day.
- Stage 3 MMF + Voclosporin: Participants receive up to 24 weeks of MMF plus 23.7 mg voclosporin (3 x 7.9 mg capsules) twice daily. Participants who previously received placebo in Stage 2 receive a scheduled ramp-up of MMF for the first two weeks.
  Participants who received placebo in Stage 2:
  * Week 1: participants receive 500 mg MMF plus matching MMF placebo (to appear like a 1000mg dose) twice daily
  * Week 2: participants receive 500 mg plus matching placebo for MMF (to appear like a 1000 mg dose) and 1000 mg MMF in divided doses
  * Weeks 3-24: 1000 mg MMF twice daily
  Participants who receive MMF in Stage 2:
  • Weeks 1-24: 1000 mg MMF twice daily
- Stage 3 MMF + Placebo for Voclosporin: Participants receive up to 24 weeks of MMF plus 23.7 mg voclosporin placebo (3 x 7.9 mg capsules) twice daily. Participants who previously received MMF placebo in Stage 2 receive a scheduled ramp-up of MMF for the first two weeks.
  Participants who received placebo in Stage 2:
  * Week 1: participants receive 500 mg MMF plus matching MMF placebo (to appear like a 1000mg dose) twice daily
  * Week 2: participants receive 500 mg plus matching placebo for MMF (to appear like a 1000 mg dose) and 1000 mg MMF in divided doses
  * Weeks 3-24: 1000 mg MMF twice daily
  Participants who received MMF in Stage 2:
  • Weeks 1-24: 1000 mg MMF twice daily
Period: Stage 2
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Started | 4 | 4 | 0 | 0
Completed (Stage 2 completion is defined as having a Stage 2 Week 48 visit.) | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 0 | 0
Not completed — Study stopped | 1 | 1 | 0 | 0
Not completed — Stage 2 Treatment Failure | 2 | 3 | 0 | 0
Not completed — Logistical issues due to participant moving | 1 | 0 | 0 | 0
Period: Stage 3
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Started | 0 | 0 | 2 | 1
Completed | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 1 | 1
Not completed — Stage 3 Treatment Failure | 0 | 0 | 0 | 1
Not completed — Study Stopped | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified Intent-to-Treat population includes all Stage 2 randomized participants who received at least one dose of Stage 2 study drug.
Groups:
- Stage 3 MMF + Placebo for Voclosporin: Participants receive up to 24 weeks of MMF plus 23.7 mg volvlosporin placebo (3 x 7.9 mg capsules) twice daily. Participants who previously received MMF placebo in Stage 2 receive a scheduled ramp-up of MMF for the first two weeks.
  Participants who received placebo in Stage 2:
  * Week 1: participants receive 500 mg MMF plus matching placebo (to appear like a 1000mg dose) twice daily
  * Week 2: participants receive 500 mg plus matching placebo for MMF (to appear like a 1000 mg dose) and 1000 mg MMF in divided doses
  * Weeks 3-24: 1000 mg MMF twice daily
  Participants who received MMF in Stage 2:
  • Weeks 1-24: 1000 mg MMF twice daily
- Total: Total of all reporting groups
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin | Total
Number analyzed (Participants) | 4 | 4 | 2 | 1 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are being reported separately for Stage 2 and Stage 3. The participants in Stage 3 are a subset of the participants in Stage 2.
  years
    Stage 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
    Stage 2 | 40.5 (15.89) | 42.5 (12.77) |  |  | 39.4 (11.16)
    Stage 3: number analyzed (Participants) | 0 | 0 | 2 | 1 | 3
    Stage 3 |  |  | 39.5 (13.44) | 53.0 (NA) — Standard deviation cannot be calculated since there is only one participant. | 44.0 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are being reported separately for Stage 2 and Stage 3. The participants in Stage 3 are a subset of the participants in Stage 2.
  Participants
    Stage 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
    Stage 2: Female | 4 | 4 |  |  | 8
    Stage 2: Male | 0 | 0 |  |  | 0
    Stage 3: number analyzed (Participants) | 0 | 0 | 2 | 1 | 3
    Stage 3: Female |  |  | 2 | 1 | 3
    Stage 3: Male |  |  | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for Stage 2 and Stage 3. The participants in Stage 3 are a subset of the participants in Stage 2.
  Participants
    Stage 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
    Stage 2: Hispanic or Latino | 0 | 1 |  |  | 1
    Stage 2: Not Hispanic or Latino | 4 | 3 |  |  | 7
    Stage 2: Unknown or Not Reported | 0 | 0 |  |  | 0
    Stage 3: number analyzed (Participants) | 0 | 0 | 2 | 1 | 3
    Stage 3: Hispanic or Latino |  |  | 0 | 0 | 0
    Stage 3: Not Hispanic or Latino |  |  | 2 | 1 | 3
    Stage 3: Unknown or Not Reported |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for Stage 2 and Stage 3. The participants in Stage 3 are a subset of the participants in Stage 2.
  Participants
    Stage 2: number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
    Stage 2: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Stage 2: Asian | 0 | 0 |  |  | 0
    Stage 2: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Stage 2: Black or African American | 1 | 1 |  |  | 2
    Stage 2: White | 3 | 2 |  |  | 5
    Stage 2: More than one race | 0 | 1 |  |  | 1
    Stage 2: Unknown or Not Reported | 0 | 0 |  |  | 0
    Stage 3: number analyzed (Participants) | 0 | 0 | 2 | 1 | 3
    Stage 3: American Indian or Alaska Native |  |  | 0 | 0 | 0
    Stage 3: Asian |  |  | 0 | 0 | 0
    Stage 3: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Stage 3: Black or African American |  |  | 0 | 0 | 0
    Stage 3: White |  |  | 1 | 1 | 2
    Stage 3: More than one race |  |  | 1 | 0 | 1
    Stage 3: Unknown or Not Reported |  |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Stage 2 Region of Enrollment Population: Data are being reported separately for Stage 2 and Stage 3. The participants in Stage 3 are a subset of the participants in Stage 2.
  participants
    United States: number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
    United States | 4 | 4 |  |  | 8
Region of Enrollment [Number; unit: participants] — Stage 3 Region of Enrollment Population: Data are being reported separately for Stage 2 and Stage 3. The participants in Stage 3 are a subset of the participants in Stage 2.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 2 | 1 | 3
    United States |  |  | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Experience a Stage 2 Treatment Failure at or Before the Stage 2 Week 24 Visit.
Description: Treatment failure is defined as the first occurrence after randomization (Stage 2) of any of the following events:
  1. Methylprednisolone acetate injection or treatment with a new or increased lupus medication, except the occasional use of corticosteroids for reasons not associated with Systemic Lupus Erythematosus (SLE) flare
  2. British Isles Lupus Assessment Group (BILAG) flare, defined as any item marked new or worse that could support a BILAG A (severe flare) or 2 organs with items marked new or worse that could support a BILAG B (moderate flare), and if the participant's condition is deemed by the investigator to be "moderately worse" or "much worse" compared to the day of randomization, as assessed by the Clinician Global Impression of Change (CGI-C)
  3. Premature permanent discontinuation of study-assigned treatment for any reason
Time Frame: From Baseline to Stage 2 Week 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF
Number analyzed (Participants) | 4 | 4
Participants | 2 | 2

2. Secondary Outcome: Clinical Response in Stage 2, Defined by the BILAG-based Combined Lupus Assessment (BICLA) at Stage 2 Week 24.
Description: The BILAG-based Composite Lupus Assessment (BICLA) is a composite index used to assess disease activity in SLE. A BICLA response is defined as meeting all of the following criteria:
  * Improvement of all Screening BILAG A scores to B, C or D
  * Improvement of all Screening BILAG B scores to C or D
  * No new BILAG A score among organs scored as B, C, D, or E at Screening
  * <= 1 new BILAG B score among organs scored as C, D, or E at Screening
  * No worsening of the Hybrid Systemic Lupus Erythematosus Disease Activity Index (H-SLEDAI)
  * Less than a 10% increase (worsening) in the Physician's Global Assessment (PGA)
  Participants who experience treatment failure prior to Stage 2 Week 24 visit are imputed as BICLA Non-responders at Stage 2 Week 24. Participants who do not have evaluable data at Stage 2 Week 24 for reasons other than a treatment failure are not imputed.
Time Frame: Stage 2 Week 24
Population: Includes all Stage 2 randomized participants who received at least one dose of Stage 2 study drug and had evaluable data at the Stage 2 Week 24 visit. Participants who experience treatment failure prior to Stage 2 Week 24 visit are considered BICLA Non-responders at Stage 2 Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF
Number analyzed (Participants) | 3 | 3
Participants
  BICLA Responder | 1 | 0
  BICLA Non-responder | 2 | 3

3. Secondary Outcome: The Proportion of Participants Who Experience a Stage 3 Treatment Failure, After Stage 3 Re-randomization at or Before Completing Stage 3 Week 24.
Description: Treatment failure is defined as the first occurrence after re-randomization (Stage 3) of any of the following events:
  1. Methylprednisolone acetate injection or treatment with a new or increased lupus medication, except the occasional use of corticosteroids for reasons not associated with Systemic Lupus Erythematosus (SLE) flare
  2. British Isles Lupus Assessment Group (BILAG) flare, defined as any item marked new or worse that could support a BILAG A (severe flare) or 2 organs with items marked new or worse that could support a BILAG B (moderate flare), and if the participant's condition is deemed by the investigator to be "moderately worse" or "much worse" compared to the day of randomization, as assessed by the Clinician Global Impression of Change (CGI-C)
  3. Premature permanent discontinuation of study-assigned treatment for any reason
Time Frame: From re-randomization to Stage 3 Week 24
Population: The Stage 3 modified Intent-to-Treat population consists of all Stage 3 re-randomized participants who received at least one dose of Stage 3 study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 3 MMF + Voclosporin: Participants receive up to 24 weeks MMF plus 23.7 mg voclosporin (3 x 7.9 mg capsules) twice daily. Participants who previously received placebo in Stage 2 receive a scheduled ramp-up of MMF for the first two weeks.
  Participants who received placebo in Stage 2:
  * Week 1: participants receive 500 mg MMF plus matching MMFplacebo (to appear like a 1000mg dose) twice daily
  * Week 2: participants receive 500 mg plus matching placebo for MMF (to appear like a 1000 mg dose) and 1000 mg MMF in divided doses
  * Weeks 3-24: 1000 mg MMF twice daily
  Participants who receive MMF in Stage 2:
  • Weeks 1-24: 1000 mg MMF twice daily
- Stage 3 MMF + Placebo for Voclosporin: Participants receive up to 24 weeks of MMF plus 23.7 mg voclosporin placebo (3 x 7.9 mg capsules) twice daily. Participants who previously received placebo in Stage 2 receive a scheduled ramp-up of MMF for the first two weeks.
  Participants who received placebo in Stage 2:
  * Week 1: participants receive 500 mg MMF plus matching MMF placebo (to appear like a 1000mg dose) twice daily
  * Week 2: participants receive 500 mg plus matching placebo for MMF (to appear like a 1000 mg dose) and 1000 mg MMF in divided doses
  * Weeks 3-24: 1000 mg MMF twice daily
  Participants who received MMF in Stage 2:
  • Weeks 1-24: 1000 mg MMF twice daily
Arm/Group | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

4. Secondary Outcome: Time to Treatment Failure in Stage 3, Defined as the Interval From the Day of Stage 3 Randomization Until the Day of Treatment Failure.
Description: as for outcome 3
Time Frame: Start of Stage 3 up to the day of treatment failure
Population: All Stage 3 re-randomized participants who received at least one dose of Stage 3 study drug and experienced a Stage 3 treatment failure.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Stage 3 MMF + Voclosporin: Participants receive up to 24 weeks MMF plus 23.7 mg voclosporin (3 x 7.9 mg capsules) twice daily. Participants who previously received placebo in Stage 2 receive a scheduled ramp-up of MMF for the first two weeks.
  Participants who received placebo in Stage 2:
  * Week 1: participants receive 500 mg MMF plus matching MMF placebo (to appear like a 1000mg dose) twice daily
  * Week 2: participants receive 500 mg plus matching placebo for MMF (to appear like a 1000 mg dose) and 1000 mg MMF in divided doses
  * Weeks 3-24: 1000 mg MMF twice daily
  Participants who receive MMF in Stage 2:
  • Weeks 1-24: 1000 mg MMF twice daily
- Stage 3 MMF + Placebo for Voclosporin: Participants receive up to 24 weeks MMF plus 23.7 mg voclosporin placebo (3 x 7.9 mg capsules) twice daily. Participants who previously received placebo in Stage 2 receive a scheduled ramp-up of MMF for the first two weeks.
  Participants who received placebo in Stage 2:
  * Week 1: participants receive 500 mg MMF plus matching MMF placebo (to appear like a 1000mg dose) twice daily
  * Week 2: participants receive 500 mg plus matching placebo for MMF (to appear like a 1000 mg dose) and 1000 mg MMF in divided doses
  * Weeks 3-24: 1000 mg MMF twice daily
  Participants who received MMF in Stage 2:
  • Weeks 1-24: 1000 mg MMF twice daily
Arm/Group | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Number analyzed (Participants) | 0 | 1
Days |  | 69 (NA) — Standard deviation cannot be calculated since there is only one participant

5. Secondary Outcome: Clinical Response in Stage 3, Defined by the BILAG-based Combined Lupus Assessment (BICLA) at Stage 3 Week 24.
Description: The BILAG-based Composite Lupus Assessment (BICLA) is a composite index used to assess disease activity in SLE. A BICLA response is defined as meeting all of the following criteria:
  * Improvement of all Screening BILAG A scores to B, C or D
  * Improvement of all Screening BILAG B scores to C or D
  * No new BILAG A score among organs scored as B, C, D, or E at Screening
  * <= 1 new BILAG B score among organs scored as C, D, or E at Screening
  * No worsening of the Hybrid Systemic Lupus Erythematosus Disease Activity Index (H-SLEDAI)
  * Less than a 10% increase (worsening) in the Physician's Global Assessment (PGA)
  Participants who experience treatment failure prior to Stage 3 Week 24 visit are imputed as BICLA Non-responders at Stage 2 Week 24. Participants who do not have evaluable data at Stage 3 Week 24 for reasons other than a treatment failure are not imputed.
Time Frame: Stage 3 Week 24
Population: Includes all Stage 3 re-randomized participants who received at least one dose Stage 3 study drug and had evaluable data at the Stage 3 Week 24 visit. Participants who experience treatment failure prior to Stage 3 Week 24 visit are considered BICLA Non-responders at Stage 3 Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Number analyzed (Participants) | 1 | 1
Participants
  BICLA Responder | 0 | 0
  BICLA Non-responder | 1 | 1

6. Secondary Outcome: The Incidence of Grade 3 or Higher Related Adverse Events (AEs) in Stage 2
Description: Defined as adverse events that emerged during Stage 2 that are of Grade 3 or higher with a relationship to Stage 2 study drug of Possible or Definite.
Time Frame: Stage 2 Day 0 up to Stage 2 Week 48
Population: Includes all participants who received at least one dose of Stage 2 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

7. Secondary Outcome: The Incidence of Grade 3 or Higher Related Adverse Events (AEs) in Stage 3
Description: Defined as adverse events that emerged during Stage 3 that are of Grade 3 or higher with a relationship to Stage 3 study drug of Possible or Definite.
Time Frame: After Stage 3 re-randomization Day 0 to Stage 3 Week 24
Population: Includes all participants who received at least one dose of Stage 3 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

8. Secondary Outcome: The Incidence of Grade 3 or Higher Infections in Stage 1
Description: Defined as infection adverse events that emerged during Stage 1 and are of Grade 3 or higher.
Time Frame: Day -28 to Day -1
Population: Includes all participants who receive at least one IM injection of a long-acting corticosteroid or who initiate withdrawal of lupus medications in Stage 1.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1: All participants who receive at least one IM injection of a long-acting corticosteroid or who initiate withdrawal of lupus medications in Stage 1
Arm/Group | Stage 1
Number analyzed (Participants) | 12
Participants | 0

9. Secondary Outcome: The Incidence of Grade 3 or Higher Infections in Stage 2
Description: Defined as infection adverse events that emerged during Stage 2 and are of Grade 3 or higher.
Time Frame: Stage 2 Day 0 up to Stage 2 Week 48
Population: Includes participants who received at least one dose of Stage 2 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF
Number analyzed (Participants) | 4 | 4
Participants | 0 | 1

10. Secondary Outcome: The Incidence of Grade 3 or Higher Infections in Stage 3
Description: Defined as infection adverse events that emerged during Stage 3 and are of Grade 3 or higher.
Time Frame: After Stage 3 re-randomization Day 0 to Stage 3 Week 24
Population: Includes participants who received at least one dose of Stage 3 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

11. Secondary Outcome: The Incidence of Renal Dysfunction in Stage 1
Description: Defined as Grade 3 or higher chronic kidney disease with eGFR < 30 ml/min per 1.73 m^2
Time Frame: Day -28 to Day -1
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1
Number analyzed (Participants) | 12
Participants | 0

12. Secondary Outcome: The Incidence of Renal Dysfunction in Stage 2
Description: Defined as Grade 3 or higher chronic kidney disease with eGFR < 30 ml/min per 1.73 m^2
Time Frame: Stage 2 Day 0 up to Stage 2 Week 48
Population: Includes participants who received at least one dose of Stage 2 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

13. Secondary Outcome: The Incidence of Renal Dysfunction in Stage 3
Description: Defined as Grade 3 or higher chronic kidney disease with eGFR < 30 ml/min per 1.73 m^2
Time Frame: After Stage 3 re-randomization Day 0 to Stage 3 Week 24
Population: Includes participants who received at least one dose Stage 3 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

14. Secondary Outcome: The Incidence of Grade 3 or Higher Hypertension in Stage 1
Description: Defined as a systolic blood pressure >= 160 mm Hg or a diastolic blood pressure of >= 100 mm Hg
Time Frame: Day -28 to Day -1
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1
Number analyzed (Participants) | 12
Participants | 0

15. Secondary Outcome: The Incidence of Grade 3 or Higher Hypertension in Stage 2
Description: Defined as a systolic blood pressure >= 160 mm Hg or a diastolic blood pressure of >= 100 mm Hg
Time Frame: Stage 2 Day 0 up to Stage 2 Week 48
Population: Includes participants who received at least one dose of Stage 2 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 MMF | Stage 2 Placebo for MMF
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

16. Secondary Outcome: The Incidence of Grade 3 or Higher Hypertension in Stage 3
Description: Defined as a systolic blood pressure >= 160 mm Hg or a diastolic blood pressure of >= 100 mm Hg
Time Frame: After Stage 3 re-randomization Day 0 to Stage 3 Week 24
Population: Includes participants who received at least one dose Stage 3 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo for Voclosporin
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs Grade 2+ or COVID-19 AEs Grade 1+ from consent until study completion, or until 30 days after early withdrawal (without withdrawing consent), or withdrawal from study, up to 56 weeks. Max time to complete Stage 2 is 4 weeks in Stage 1 + 48 weeks in Stage 2 + 4 weeks in Safety F/U = 56 weeks. For Stage 3, treatment failure occurs at or before Stage 2 Week 24 visit. Max time to complete Stage 3 is 4 weeks in Stage 1 + 24 weeks in Stage 2 + 24 weeks in Stage 3 +4 weeks in Safety F/U = 56 weeks.
Description: AEs are reported in the stage in which the event emerged
Groups:
- Stage 1 Corticosteroid During Treatment Withdrawal: Participants receive up to 3 corticosteroid injections to achieve amelioration of symptoms and withdraw from lupus treatments. Stage 1 may last up to 4 weeks.
- Stage 2 MMF: Participants receive 1000 mg MMF twice daily (following a 2 week ramp up) for up to 48 weeks.
- Stage 2 Placebo: Participants receive Placebo twice daily for up to 48 weeks.
- Stage 3 MMF + Voclosporin: Participants receive 1000 mg MMF twice daily (following a 2 week ramp up) plus 23.7 mg of Voclosporin twice daily for up to 24 weeks.
- Stage 3 MMF + Placebo: Participants receive 1000 mg MMF twice daily (following a 2 week ramp up) plus Placebo twice daily for up to 24 weeks.
Arm/Group | Stage 1 Corticosteroid During Treatment Withdrawal | Stage 2 MMF | Stage 2 Placebo | Stage 3 MMF + Voclosporin | Stage 3 MMF + Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 1/4 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/12 | 3/4 | 3/4 | 1/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Corticosteroid During Treatment Withdrawal (N=12) | Stage 2 MMF (N=4) | Stage 2 Placebo (N=4) | Stage 3 MMF + Voclosporin (N=2) | Stage 3 MMF + Placebo (N=1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Corticosteroid During Treatment Withdrawal (N=12) | Stage 2 MMF (N=4) | Stage 2 Placebo (N=4) | Stage 3 MMF + Voclosporin (N=2) | Stage 3 MMF + Placebo (N=1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT05306873/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05306873/ICF_000.pdf